CLINICAL TRIAL: NCT01286805
Title: Lumbar Plexus Block for Postoperative Pain Control After Hip Arthroscopy. A Randomized Controlled Trial
Acronym: LPB Hip Scope
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: New York Presbyterian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10038
Record Dates: First submitted 2011-01-28; First posted 2011-01-31 (Estimated); Results first posted 2013-06-05 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-05

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lumbar Plexus Blockade + CSE (Experimental): The study group will receive a lumbar plexus blockade with 30 mL of 0.25% bupivacaine with 1:200,000 epinephrine, followed by a combined spinal-epidural.
  Interventions: Procedure: Lumbar Plexus Blockade
- Control Group (Placebo Comparator): The control group will receive only a combined spinal-epidural.
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Lumbar Plexus Blockade — The lumbar plexus block will be dosed with 30 milliliters of 0.25% bupivacaine with 1:200,000 epinephrine
  Other Names: Marcaine
  Arms: Lumbar Plexus Blockade + CSE
Procedure: Control — The control group will receive only a combined spinal-epidural.
  Arms: Control Group

SUMMARY:
The purpose of this study is to determine whether the use of a lumbar plexus block for arthroscopic hip surgery is superior to oral and intravenous opioid pain medications alone in treating pain. In addition, the study will examine whether lumbar plexus blocks reduce the total amount of pain medication needed, and therefore reduce the side effects of these medicines and increase patient satisfaction. It is hypothesized that addition of the lumbar plexus block will significantly reduce patients' postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Class 1-3
* Patients aged 18 to 65 years
* Patients scheduled for primary, unilateral arthroscopic hip surgery by Dr. Kelly, Dr. Coleman, or Dr. Anil Ranawat
* Planned use of neuraxial anesthesia
* Body Mass Index less than 35
* Ability to follow study protocol

Exclusion Criteria:

* Chronic opioid use (defined as daily or almost daily use of opioids for >3 months)
* Contraindication to combined spinal-epidural anesthesia including but not limited to bleeding disorder, use of clinically relevant anticoagulant or antiplatelet medications, and anatomic abnormalities.
* Contraindication to lumbar plexus block including but not limited to bleeding disorder, use of clinically relevant anticoagulant or antiplatelet medications, and anatomic abnormalities.
* Infection at the injection site(s)
* Allergy to any of the study medications
* Contraindication to a short course of NSAIDs (renal failure, intolerance)
* ASA Class 4-5
* Patient refusal
* Patients younger than 18 years old and older than 65
* Patients with any known indwelling hardware of the lumbar spine.
* Patients with a peripheral neuropathy of the surgical extremity
* Non-English speaking patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2010-05; Primary Completion 2010-10 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques T YaDeau, M.D., Ph.D., Principal Investigator — Hospital for Special Surgery, New York
Locations (2):
- United States (2):
  - Hospital for Special Surgery, New York, New York
  - New York Presbyterian Hospital, New York, New York

REFERENCES:
- See also: This is the link for the Hospital for Special Surgery website — http://www.hss.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Lumbar Plexus Blockade + CSE: The study group received a lumbar plexus blockade with 30 mL of 0.25% bupivacaine with 1:200,000 epinephrine, followed by a combined spinal-epidural.
- Control Group: The control group received only a combined spinal-epidural.
Period: Overall Study
Arm/Group | Lumbar Plexus Blockade + CSE | Control Group
Started | 41 | 42
Completed | 41 | 41
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lumbar Plexus Blockade + CSE | Control Group | Total
Number analyzed (Participants) | 41 | 41 | 82
Age Continuous [Mean (Standard Deviation); unit: years] | 33 (11) | 37 (11) | 35 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 20 | 21 | 41

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Scale (NRS) Pain at Rest (0-10) on Day of Surgery Prior to Discharge
Description: The Numeric Rating Scale was used to ask patients to rate their pain at rest on a scale of 0 to 10, 0 = no pain and 10 = worst pain imaginable.
Time Frame: Day of surgery prior to discharge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lumbar Plexus Blockade + CSE | Control Group
Number analyzed (Participants) | 41 | 41
units on a scale | 3.3 (2.2) | 4.2 (1.8)

2. Secondary Outcome: Readiness to Discharge From Post-Anesthesia Care Unit (PACU)
Description: Time to readiness for discharge from the PACU. Patients were considered ready for PACU discharge when they met the following criteria: a) Awake, alert, oriented and responsive b) Minimal pain, Numeric Rating Scale < 5/10 (0 = no pain, 10 = worst imaginable pain) (parenteral [injected] medications not required) c) Vital signs stable d) No active bleeding e) Minimal or no nausea f) Not vomiting, tolerating oral intake g) Oxygen saturation > 94% (or baseline) on room air h) Patient has urinated.
Time Frame: Day of surgery prior to discharge
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Lumbar Plexus Blockade + CSE | Control Group
Number analyzed (Participants) | 41 | 41
minutes | 216 (86) | 187 (59)

3. Secondary Outcome: Narcotic Pain Medication Needed
Time Frame: Day of surgery prior to discharge
Measure: Mean (Standard Deviation); unit: equivalents milligrams oral morphine
Arm/Group | Lumbar Plexus Blockade + CSE | Control Group
Number analyzed (Participants) | 41 | 41
equivalents milligrams oral morphine | 21 (17) | 29 (21)

4. Secondary Outcome: Incidence of Nausea
Description: The number of participants with nausea.
Time Frame: Day of surgery prior to discharge
Measure: Number; unit: participants
Arm/Group | Lumbar Plexus Blockade + CSE | Control Group
Number analyzed (Participants) | 41 | 41
participants | 14 | 8

5. Secondary Outcome: Incidence of Vomiting
Description: The number of participants who vomited.
Time Frame: Day of surgery prior to discharge
Measure: Number; unit: participants
Arm/Group | Lumbar Plexus Blockade + CSE | Control Group
Number analyzed (Participants) | 41 | 41
participants | 1 | 3

6. Secondary Outcome: Requirement of Antiemetic Rescue
Description: The number of participants who needed medication to treat their nausea and vomiting.
Time Frame: Day of surgery prior to discharge
Measure: Number; unit: participants
Arm/Group | Lumbar Plexus Blockade + CSE | Control Group
Number analyzed (Participants) | 41 | 41
participants | 5 | 5

7. Secondary Outcome: Patient Satisfaction
Description: Patient Satisfaction (0-10; 0 = very dissatisfied, 10 = very satisfied)
Time Frame: First 24 hours after surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lumbar Plexus Blockade + CSE | Control Group
Number analyzed (Participants) | 41 | 41
units on a scale | 8.6 (1.6) | 7.9 (2.5)

8. Secondary Outcome: Quality of Recovery (QoR-40) Physical Comfort Dimension
Description: Assessment of Physical Comfort (minimum score = 12, maximum score = 60). Higher values represent a better outcome
Time Frame: First 24 hours after surgery
Measure: Mean (Standard Deviation); unit: QoR-40 Physical Comfort score
Arm/Group | Lumbar Plexus Blockade + CSE | Control Group
Number analyzed (Participants) | 41 | 41
QoR-40 Physical Comfort score | 53 (4.3) | 52 (7.4)

ADVERSE EVENTS:
Arm/Group | Lumbar Plexus Blockade + CSE | Control Group
Serious Adverse Events (participants affected / at risk) | 3/42 | 2/41
Other Adverse Events (participants affected / at risk) | 0/42 | 0/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lumbar Plexus Blockade + CSE (N=42) | Control Group (N=41)
Admission for nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) — 1 control patient was admitted to the hospital for intractable nausea (attributed to opioid analgesics)
Admission for oxygen desaturation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — 1 control patient was admitted to the hospital for hypoxemia (attributed to opioid analgesics)
Fall (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) — 2 LPB patients fell in the hospital bathroom without injury
Admission for epidural spread (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — 1 LPB patient was admitted for epidural spread and urinary retention (procedural complication)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes